CLINICAL TRIAL: NCT03343288
Title: The Use of Silver Doped Calcium Phosphate Based Ceramic Coated Orthopedic Implants for Preventing Implant Related Infection
Brief Title: Silver Doped Ceramic Coated Orthopedic Implants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, NUSRET KOSE, Professor of Orhopedics and Traumatology, Eskisehir Osmangazi University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 315S101
Record Dates: First submitted 2017-10-22; First posted 2017-11-17 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Implant Site Infection; Implant Infection
Keywords: Silver Hydroxiapatite Coating; Antimicrobial; Medical Device

STUDY DESIGN:
Intervention Model Description: In this study, hip joint prostheses, intramedullary nails and external fixator implants to be used in 30 patients . CE marked, domestic manufactured standard orthopedic implants will be used in patients after silver doped HA coating . Antimicrobial effectiveness of the coating will be evaluated. These patients will be tasted for the evaluation of liver and kidney functions and blood and urine silver levels in addition to routine tests such as full blood, complete biochemistry, C-reactive protein, erythrocyte sedimentation rate required in the normal diagnosis and treatment processes, and will be monitored for at least 12 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Silver HA coated implants (Experimental): Silver doped hydroxyapatite coated implants
  Interventions: Device: Silver doped hydroxyapatite coated implants

INTERVENTIONS:
Device: Silver doped hydroxyapatite coated implants — In this study, CE marked, domestic manufactured standard orthopedic implants will be used in 30 patients after silver ceramic coating with electrospray method. These patients will be tasted for the evaluation of liver and kidney functions and blood and urine silver levels in addition to routine tests such as full blood, complete biochemistry, C-reactive protein, erythrocyte sedimentation rate required in the normal diagnosis and treatment processes, and will be monitored for at least 12 months.

SUMMARY:
In this study, CE (European Conformity) marked, domestic manufactured standard orthopedic implants will be used after silver HA coating with electrospray method in 30 patients requiring hip joint prostheses, intramedullary nails or external fixator in 30 patients to antimicrobial effectiveness. These patients will be tasted for liver and kidney functions and blood and urine silver levels in addition to routine tests such as full blood, complete biochemistry, C-reactive protein, erythrocyte sedimentation rate required in the normal diagnosis and treatment processes,

DETAILED DESCRIPTION:
In this study, considering the differences in bone contact surface area and interactions; hip joint prostheses, intramedullary nails and external fixator implants to be used in 30 patients . CE (European Conformity) marked, domestic manufactured standard orthopedic implants will be used in patients after silver HA coating with electrospray method. These patients will be tasted for the evaluation of liver and kidney functions and blood and urine silver levels in addition to routine tests such as full blood, complete biochemistry, C-reactive protein, erythrocyte sedimentation rate required in the normal diagnosis and treatment processes, and will be monitored for at least 12 months. The performance of coating to be applied and any unwanted side effects in normal conditions of use will be evaluated..

ELIGIBILITY:
Inclusion Criteria:

1. Men and women between the ages of 18-65
2. Patients without heart, lung, renal or hepatic insufficiency
3. Patients without epilepsy, cerebrovascular attack or ischaemia
4. Patients without antibiotic allergy
5. Patients who have low immune defense mechanisms such as malignancy, diabetes mellitus, polytrauma, and open fracture
6. Patients using oral or parenteral corticosteroids, methotrexate, cyclosporine or other immunosuppressive drugs - -

Exclusion Criteria:

1. Pregnant women
2. Patients with another silver implant in their body, such as a silver-coated stent
3. Patients with known allergy or hypersensitivity to silver
4. Patients with too many antibiotics due to recurrent infections

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Number of pin site with positive culture resuls | 12 months
  incidence of pin tract infection

SECONDARY OUTCOMES:
Number of patient with elevated level of serum ALT levels | 12 months
  liver dysfunction
Number of patient with elevated BUN levels | 12 months
  Kidney dysfunction
Number of patient with elevated blood silver | 12 months
  Silver exposure

CONTACTS AND LOCATIONS:
Overall Officials: Nusret kose, MD, Principal Investigator — Eskisehir Osmangazi University
Locations (1):
- Eskisehir Osmangazi University Hospital, Eskişehir, Turkey (Türkiye)